CLINICAL TRIAL: NCT02097927
Title: The Effect of Sensory-enhanced Beverages on Satiety Following Repeated Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leatherhead Food Research (Industry)
Collaborators: University of Sussex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 127438-1
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Subjects
Keywords: Appetite; Satiety; Energy intake; Saliva; Biomarkers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- High energy, low sensory (Experimental): Mango-flavour beverage
  Interventions: Behavioral: Mango-flavour beverage
- Low energy, high sensory (Experimental): Mango-flavour beverage
  Interventions: Behavioral: Mango-flavour beverage
- High energy, high sensory beverage (Experimental): Mango-flavour beverage
  Interventions: Behavioral: Mango-flavour beverage

INTERVENTIONS:
Behavioral: Mango-flavour beverage — The study will be a 3-way crossover design: it will assess the impact of a high-energy, sensory-enhanced beverage on energy intake through ad libitum food consumption and subjective feeling of appetite using visual analogue scales (VAS) compared to 2 control beverages following repeated exposures. Each participant will consume each beverage 10 times. This includes 2 satiety-testing sessions on site at Leatherhead Food Research, and 8 occasions consuming the product as a mid-morning snack during the participants' normal routine. Each participant will attend the Nutrition Unit on 6 different occasions before and after repeated exposures to the beverages at home. There will be a two-week washout period in which none of the beverages are consumed between the different beverage manipulations.

SUMMARY:
The study will be a 3-way crossover design: it will assess the impact of consuming a beverage enhanced with satiety-relevant properties on subjective ratings of appetite and on energy intake compared with a low energy version with the same sensory characteristics, and a non-sensory enhanced high energy control.

In addition, saliva samples will be collected at regular intervals for the identification of novel biomarkers of energy intake.

DETAILED DESCRIPTION:
The study will be a 3-way crossover design: it will assess the impact of a high-energy, sensory-enhanced beverage on energy intake through ad libitum food consumption and subjective feeling of appetite using visual analogue scales (VAS) compared to 2 control beverages following repeated exposures. Each participant will consume each beverage 10 times. This includes 2 satiety-testing sessions on site at Leatherhead Food Research, and 8 occasions consuming the product as a mid-morning snack during the participants' normal routine. Each participant will attend the Nutrition Unit on 6 different occasions (plus one screening visit) before and after repeated exposures to the beverages at home. The order in which participants receive the beverages will be counterbalanced and randomised. There will be a two-week washout period in which none of the beverages are consumed between the different beverage manipulations. Participants will fast overnight before each visit and consume the same evening meal before each test day. Participants will be instructed to avoid consuming food or calorific beverages for one hour before or after consuming the beverage. Following the last satiety testing day participants will be debriefed and open questions will be asked about experiences of the beverages in a focus group format.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* Age at start of the study ≥ 18 and ≤ 65 years
* Body Mass Index (BMI) ≥ 18 and ≤ 29.9 kg/m2
* Apparently healthy: measured by questionnaire (APPENDIX 3): no reported current or previous metabolic diseases or chronic gastrointestinal disorders
* Reported dietary habits: no medically prescribed diet, no slimming diet, used to eating 3 meals a day
* Reported intense sporting activities ≤ 10h/w
* Reported alcohol consumption ≤14 units/w
* Informed consent signed
* Recruitment form filled out

Exclusion Criteria:

* Smoking
* Dislike, allergy or intolerance to test products or study meals
* Possible eating disorder (measured by SCOFF questionnaire score >1)
* Reported medical treatment that may affect eating habits/satiety
* Eating habits questionnaire score >14
* Reported participation in another biomedical trial 1 month before the start of the study
* Food allergies or intolerance to ad libitum meals
* Pregnant and/or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in energy intake | Weeks 0,3,5,8,10 and 13
  Change in intake (kcals) at an ad libitum lunch, assessed before and after the repeated exposure period for each of the 3 beverage products

SECONDARY OUTCOMES:
Change in subjective appetite ratings | Weeks 0,3,5,8,10 and 13
  Change in subjective feelings of appetite assessed with Visual Analogue Scales (VAS). These will be measured on each of the 6 test days, which will occur before and after the repeated exposure period for each of the 3 beverage products.

OTHER OUTCOMES:
Biomarkers of appetite in saliva samples | Weeks 0,3,5,8,10 and 13
  Frozen saliva samples will be banked. On completion of the study saliva samples associating with the extremes of appetite rating or energy intake will be pooled (6-12 samples / pool) and the protein component analysed by quantitative proteomics using an isobaric tags for relative and absolute quantitation (iTRAQ) workflow. Remaining samples will be retained for validation of proteins found to associate or predict appetite or energy intake.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Re, PhD, Study Director — Leatherhead Food Research
Locations (1):
- Leatherhead Food Research Nutrition Unit, Leatherhead, Surrey, United Kingdom